CLINICAL TRIAL: NCT02629341
Title: Functional Yogurt Powder Effect on Bone Health Biomarkers
Acronym: bonefoods
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Instituto de Investigación Hospital Universitario La Paz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BONEFOODS
Record Dates: First submitted 2015-12-10; First posted 2015-12-14 (Estimated); Last update posted 2015-12-14 (Estimated); Status verified 2015-12

CONDITIONS: OSTEOPENIA
Keywords: woman osteopenia osteoporosis enriched calcium vit D yogurt
MeSH Terms: conditions — Bone Diseases, Metabolic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Functional yogurt powder (Active Comparator): This arm will receive one daily serving of the functional yogurt which is enriched in Calcium, D, K, C vitamins, Zn, Mg, L-leucin and the Lactobacillus plantarum 3547 probiotic
  Interventions: Dietary Supplement: Functional yogurt powder
- Control yogurt powder (Placebo Comparator): This arm will receive one daily serving of the control yogurt which consists of a regular yogurt not enriched
  Interventions: Dietary Supplement: Control yogurt powder

INTERVENTIONS:
Dietary Supplement: Functional yogurt powder — Once daily during 24 weeks, 150g of yogurt powder enriched with:
  Calcium (mg) 501 D3 Vitamin (Colecalciferol) (μg(UI)) 6(240) K Vitamin (μg) 80 C Vitamin (mg) 100 Zinc (mg) 10,39 Magnesium (mg) 250,5 L-Leucin (g) 1 Lactobacillus plantarum 3547 (ufc) 1x10e10
  Arms: Functional yogurt powder
Dietary Supplement: Control yogurt powder — Once daily during 24 weeks, 150g of yogurt powder not enriched, isocaloric and with an equal macronutrient composition than the functional yogurt
  Arms: Control yogurt powder

SUMMARY:
The purpose of this study was to evaluate the therapeutic effect of a functional yogurt powder on menopausal, middle-aged women at high risk of osteoporosis. The functional yogurt powder containing Calcium, D, K, C vitamins, Zn, Mg, L-leucin and the Lactobacillus plantarum 3547 probiotic, was developed to benefit bone health and in the long term may contribute to the prevention of osteoporosis.

DETAILED DESCRIPTION:
Randomized, parallel, double-blind, placebo controlled clinical trial to evaluate the effect of a functional yogurt powder on bone health biomarkers in menopause, middle-aged women at high risk of osteoporosis.

78 volunteers will be recruited at the La Paz University Hospital of Madrid. Participants should meet the next inclusion criteria: being menopausal, aged between 50 and 65 years, IMC≥18.5 <35 Kg/m2 and having a diagnosis of osteopenia without pharmacological treatment (Volunteers without osteopenia diagnosis should meet two of the next: dairy intake under 2 servings a day, sedentary lifestyle and/or smokers of more than 5 cigarettes a day).

Participants will be randomized in two arms:

1. Functional yogurt powder arm: they will receive over 24 weeks a daily serving of the functional yogurt powder containing Calcium, D, K, C vitamins, Zn, Mg, L-leucin and the Lactobacillus plantarum 3547 probiotic.
2. Control yogurt powder arm: they will receive over 24 weeks a daily serving of the control yogurt powder (not enriched).

All participants will be advised to follow a healthy diet and practice physical activity.

Follow up will include 3 individualized visits and 4 group visits to check the product intake compliance and the tolerance to the product. The primary outcome, vitamin D level, will be measured at the beginning (basal condition) and at the end of the intervention (24 weeks). Other bone health biomarkers (Parathyroid hormone (PTH) calcium, phosphorus, calcitonin, osteocalcin, adrenocorticotropic hormone (ACTH),osteopontin, osteoprotegerin, sclerostin,the N-terminal telopeptide (NTx) and C-terminal telopeptide CTx) and safety issues (transaminases and creatinine) will be measured at the same time points (0 and 24 weeks).

ELIGIBILITY:
Inclusion Criteria:

* With healthy weight, overweight or obesity type I (IMC ≥18.5 <35 Kg/m2);
* With diagnosis of osteopenia without pharmacological treatment or that meet at least two of the following criteria:

  * Dairy intake under 2 servings daily in the last year
  * Sedentary lifestyle (measured with the International physical activity questionary IPAQ)
  * Smokers of more than 5 cigarettes daily
* Signed informed consent.

Exclusion Criteria:

* Severe diseases (hepatic, kidney, cancer…)
* Renal failure (defined as serum creatinine level >200 mol/L)
* Phosphate binding antacids (> 6 months a year)
* Oral glucocorticoids (>5 mg/day of prednison equivalent in the last 8 months or a total dose of 2g of prednison equivalent in the last 12 months)
* Local treatment with injectable glucocorticoids (>5 injections/year)
* Treatment with inhaled glucocorticoids (>6months in the last year and more than 2 mg/day of prednison equivalent)
* Previous or concomitant treatment for metabolic bone disease
* Use of hormone replacement therapy (oral estrogen, estradiol vaginal ring, antiestrogen, progesterone)
* Anabolic steroid use in the last 3 months or more than one in the last 6 months
* Estradiol implants in the last 3 years
* Isoflavan use in the last 6 months or more than once a month for the last 12 months
* Calcitonin use in the last month or more than 1 month in the last 6 months
* Concomitant use of nutritional supplements with silicon, horsetail extracts, bamboo, colloidal silicic acid or silanol derivatives in the last 6 months
* Hyperparathyroidism and/or hyperthyroidism
* Chronic intestinal disease (Gastritis, ulcerative colitis, irritable bowel disease, pseudomembranous colitis, inflammatory bowel disease, Crohn disease, etc)
* Dementia, mental disease or diminished cognitive function
* Mayor surgery in the last month or gastrointestinal surgery in the last 3 months
* Prebiotic, probiotic ad/or symbiotic consumption, antioxidant supplements, supplements with omega 3, vitamins or minerals in the last 2 weeks prior to the start of the study
* Participation in programs and / or drug use for weight control in the last 6 months
* Alcohol consumption over 30g/day
* Habitual laxative use and non acceptance in giving up its use during the study

  * Individuals using topic glucocorticoids can enter the trial

Ages: 50 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2015-01; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
changes in plasma 25(OH)D concentration | 0 and 24 weeks

SECONDARY OUTCOMES:
Change from baseline Body composition by Dual-energy X-ray absorptiometry (DXA) | 0 and 24 weeks
Change from baseline calcium levels in blood | 0 and 24 weeks
Change from baseline Parathyroid hormone (PTH) | 0 and 24 weeks
Change from baseline adrenocorticotropic hormone (ACTH) | 0 and 24 weeks
Change from baseline Calcitonin | 0 and 24 weeks
Change from baseline osteocalcin | 0 and 24 weeks
Change from baseline Osteopontin | 0 and 24 weeks
Change from baseline Osteoprotegerin | 0 and 24 weeks
Change from baseline sclerostin | 0 and 24 weeks
Change from baseline phosphorus | 0 and 24 weeks
Change from baseline N-terminal telopeptide | 0 and 24 weeks
Change from baseline the C-terminal telopeptide | 0 and 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Gomez Candela, MD, PhD, Principal Investigator — Hospital Universitario La Paz
Locations (1):
- Hospital Universitairo La Paz, Madrid, Madrid, Spain